CLINICAL TRIAL: NCT00756951
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Dose Ranging Study to Assess the Safety and Efficacy of SC-07 for the Delay to Onset of Severe Oral Mucositis in Subjects Receiving Chemoradiation Therapy for the Treatment of Cancers of the Head and Neck.
Brief Title: Dose Ranging Study to Assess the Safety and Efficacy of SCV-07 for the Delay to Onset of Severe Oral Mucositis in Patients Receiving Chemoradiation Therapy for Head and Neck Cancer
Acronym: SCV-07 OM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Israel Rios, MD, SciClone Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: SCI-SCV-MUC-P2-001
Record Dates: First submitted 2008-09-12; First posted 2008-09-22 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2008-12

CONDITIONS: Oral Mucositis; Head and Neck Cancer
Keywords: SCV-07; Oral Mucositis
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms | interventions — golotimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Active Comparator): SCV-07 at a dose of 0.02 mg/kg
  Interventions: Drug: SCV-07
- 3 (Active Comparator): SCV-07 at a dose of 0.10 mg/kg
  Interventions: Drug: SCV-07

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: 1
Drug: SCV-07 — 0.02 mg/kg
  Arms: 2
Drug: SCV-07 — 0.10 mg/kg
  Arms: 3

SUMMARY:
Oral Mucositis (OM) is a painful and debilitating side effect of many of the drug or radiation regiments used to treat cancer. This study examines the investigational drug SCV-07 and it's possible application in treating Oral Mucositis. Studies have shown that SCV-07 can possibly increase a broad immune system response, thus lowering the painful side effects experienced when treated for head and neck cancer.

The purpose of this study is to assess the safety and tolerability of SCV-07 and it's ability to delay the onset of Oral Mucositis for patients receiving chemoradiation for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a body weight less than 150 kg at screening
* Have recently-diagnosed, pathologically-confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx that will be treated with chemoradiation therapy as first line treatment(postoperative patients are eligible, if surgery is < 6 weeks prior to initiation of radiotherapy.
* Plan to receive a continuous course of conventional external beam irradiation
* Plan to receive a standard cisplatin chemotherapy regimen

Exclusion Criteria:

* Pregnant or breastfeeding
* Have head and neck tumors of the lips, sinuses, salivary glands or unknown primary tumor
* Prior radiation to the head and neck
* Have a plan to receive cetuximab (Erbitux) in conjunction with chemotherapy
* Had curative surgery more than 6 weeks prior to the initiation of radiotherapy
* Have current oral mucositis
* Presence of active infectious disease excluding oral candidiasis
* Chronic immunosuppression
* Seropositive for HIV or hepatitis B surface antigen or C antibody
* Used an investigational agent within 30 days of randomization
* Have a known sensitivity to any investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59
Dates: Start 2008-09

PRIMARY OUTCOMES:
Safety will be assessed by collecting and recording AEs and laboratory assessments. Labs will be collected at screening,weekly throughout the subject's RT treatment and on the last day of radiotherapy. | 7 Weeks
Efficacy of Oral Mucositis assessment will be completed by trained site personnel. The WHO score will be the primary measure and NCI CTCAE will be a secondary measure for assessing Oral Mucositis. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Israel Rios, MD, Study Director — SciClone Pharmaceuticals
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Whittingham Cancer Center, Norwalk, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - University of Illinois at Chicago, Chicago, Illinois
  - James Graham Brown Cancer Center, Lousiville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St Louis, St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Beth Israel Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Ohio State University Medical Center, Columbis, Ohio
  - St Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Related Info — http://www.sciclone.com